CLINICAL TRIAL: NCT00350194
Title: Pilot Study: The Effects of Omega-3 Fatty Acids on Metabolic Syndrome and Vascular Structure in Metabolic Syndrome as Assessed by Carotid IMT
Brief Title: The Effects of Omega-3 Fatty Acids on Metabolic Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Pfizer (Industry); National Institutes of Health (NIH) (NIH); Northwest Lipid Research Clinic (Unknown)
Responsible Party: Principal Investigator, Pathmaja Paramsothy, Assistant Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 28791-D; 05-8693-D 03
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Metabolic Syndrome X
Keywords: Fatty Acids, Omega-3
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Placebo Comparator): Omega-3 fatty acid vs. placebo comparator
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — Total of 1.8 grams of EPA +DHA in the form of fish oil capsules (3/day)
  Other Names: Fish Oil

SUMMARY:
The purpose of this study is to determine the effects of omega-3 fatty acids in the form of fish oil supplementation (approximately 2 grams per day) on the carotid intima-media (CIMT)progression (primary objective) and 2)(Secondary objective) lipid markers such as LDL, apo-B, and LDL buoyancy, on inflammatory burden as measured by CRP, on oxidative stress as measured by urinary isoprostanes, urine microalbumin/creatinine, and serum adiponectin a fat derived hormone in subjects with metabolic syndrome.

DETAILED DESCRIPTION:
This translational pilot study will have a double-blind, placebo-controlled, parallel design. We will enroll one hundred subjects who meet at least 3 of the 5 criteria for metabolic syndrome as per NCEP guidelines/WHO guidelines and who do not have known cardiovascular disease or diabetes. They will receive either placebo or omega-3 fatty acids in the form of fish oil capsules for a two-year period. Assessment of, C-IMT, serum lipoprotein profile, LDL- buoyancy, adiponectin, CRP, SAA, apolipoprotein B and A-1, fasting glucose, fasting insulin levels, and plasma fatty acids will be measured at baseline, one year, and two years.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Metabolic Syndrome (meets 3 of the following 5)
* Abdominal obesity, waist circumference in men greater than 40 in. & in women greater than 35 in.
* Serum triglycerides greater than or = 150 mg/dL (1.7 mmol/L)
* Serum HDL cholesterol less than or = 40 mg/dL in men and less than 50 mg/dL in women
* Blood pressure greater than or = 130/85 mmHg or drug treatment for elevated blood pressure
* Fasting plasma glucose greater than 100 mg/dL

Exclusion Criteria:

* Diabetes
* Known or documented CHD (including ECG consistent with prior MI), CVA (including TIA), PVD (including symptoms of claudication)
* Angina or other chest pain that may indicate CHD
* Clinically significant neoplastic, cardiovascular, hepatic, renal, metabolic, endocrine (untreated or unstable), or psychiatric (untreated or unstable)
* Known abnormal LFTS greater than 2X ULN
* Smoker, illicit drug use, or excessive alcohol use
* Medications: Lipid lowering therapy, daily NSAID or greater than 325 mg ASA (PRN use ok), clopidogrel (or equivalent), Coumadin, Omega-3 fatty acid supplement, other investigational drugs within 30 days of study entry, high omega-3 fatty acid content in diet within past three months
* Pregnancy or planning pregnancy during the study period
* Sensitivity or allergy to fish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change in Carotid IMT | 1 year, 2 years

SECONDARY OUTCOMES:
Lipid (apolipoproteins and lipid parameters) | 1 year, 2 years
hs-CRP & SAA | 1 year, 2 years
Glucose | 1 year, 2 years
Insulin | 1 year, 2 years
adiponectin | 1 year, 2 years
urine microalbumin/creatinine | 1 year, 2 years
Serum Fatty Acids | 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pathmaja Paramsothy, MD, Principal Investigator — University of Washington
Locations (1):
- Northwest Lipid Research Clinic (University of Washington Affiliated), Seattle, Washington, United States